CLINICAL TRIAL: NCT02346903
Title: Chest Pain Perception and Capsaicin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, Dhananjai Menzies, MD, Attending Physician - Cardiology, Bassett Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1029
Record Dates: First submitted 2014-12-16; First posted 2015-01-27 (Estimated); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac Catheterization Patients (Other): Subjects will undergo the cutaneous capsaicin test. A one inch ribbon of Capzasin-HP Cream (0.1%) will be applied to the skin on the forearm of the non-dominant arm. Subjects will be asked to assign a numerical score to the maximum intensity of any cutaneous discomfort experienced during the subsequent 30 minutes, ranging from 0 ("no discomfort") to 10 ("the worst discomfort imaginable"). The cream will then be removed by washing the affected arm with cold water. The patients will be asked follow-up questions concerning their experiences with chest pain in the past and their tolerance of spicy foods. Efforts will then be made to examine the association between the pain score documented in response to the cutaneous capsaicin test with the pain score obtained during coronary balloon occlusion.
  Interventions: Drug: Capsaicin

INTERVENTIONS:
Drug: Capsaicin — one inch ribbon of Capzasin -HP applied to forearm for 30 minutes
  Other Names: Capzasin-HP 0.1%

SUMMARY:
The purpose of this study is to determine whether there is a positive correlation between the ability to sense chest pain in the context of myocardial ischemia and the ability to sense discomfort associated with the topical application of the TRPV1 agonist capsaicin (the active ingredient on hot chili peppers). Patients undergoing clinical elective balloon angioplasty of a coronary stenosis will be asked to quantify the subjective intensity of any chest pain they feel during a standardized episode of myocardial ischemia produced by a one-minute coronary balloon occlusion, using a previously-validated numeric rating scale. The same patients will subsequently be asked to grade the subjective intensity of cutaneous discomfort resulting from application of a capsaicin-containing patch (Capzasin-HP Cream, an over-the-counter product approved for topical application to treat muscle and joint aches) to the forearm. The goal will be to determine whether an association can be demonstrated between the subjective perception of ischemic chest pain during coronary balloon occlusion and cutaneous capsaicin sensitivity. Such an association could have considerable clinical value, as it might allow physicians to prospectively assess an individual's ability to perceive myocardial ischemia/infarction by assessing his/her subjective response to the topical application of capsaicin.

DETAILED DESCRIPTION:
Chest discomfort is considered the hallmark of myocardial ischemia and as such is an important clinical warning sign of myocardial infarction (MI). The ability to sense ischemic chest discomfort appears to be impaired in a substantial minority of the population and such individuals are presumably at increased risk for unrecognized MI. While the mechanism(s) responsible for the perception of chest pain associated with myocardial ischemia are still not fully understood, studies suggest that the transient receptor potential vanilloid-1 (TRPV1) plays a key role in this process. This nociceptor, which is known to mediate pain sensation in the skin and elsewhere in the peripheral nervous system, has also been found on the outer surface of the heart and has been shown to respond to ischemic stress in this organ.

The purpose of this study is to determine whether there is a positive correlation between the ability to sense chest pain in the context of myocardial ischemia and the ability to sense discomfort associated with the topical application of the TRPV1 agonist capsaicin (the active ingredient on hot chili peppers). Patients undergoing clinical elective balloon angioplasty of a coronary stenosis will be asked to quantify the subjective intensity of any chest pain they feel during a standardized episode of myocardial ischemia produced by a one-minute coronary balloon occlusion, using a previously-validated numeric rating scale. The same patients will subsequently be asked to grade the subjective intensity of cutaneous discomfort resulting from application of a capsaicin-containing patch (Capzasin-HP Cream, an over-the-counter product approved for topical application to treat muscle and joint aches) to the forearm. The goal will be to determine whether an association can be demonstrated between the subjective perception of ischemic chest pain during coronary balloon occlusion and cutaneous capsaicin sensitivity. Such an association could have considerable clinical value, as it might allow physicians to prospectively assess an individual's ability to perceive myocardial ischemia/infarction by assessing his/her subjective response to the topical application of capsaicin.

ELIGIBILITY:
Inclusion Criteria:

Subjects will consist of patients who have undergone clinically-indicated percutaneous coronary intervention (PCI) for the treatment of coronary artery disease.

Exclusion Criteria:

Clinically unstable patients, such as those undergoing emergency PCI, patients with documented hypersensitivity to capsaicin will be excluded and patients who have used a capsaicin-based product within the last 3 months will be excluded. Patients in whom it would be inadvisable for any reason to conduct a one-hour research study at a follow-up visit after PCI will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhananjai Menzies, MD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardiac Catheterization Patients
Started | 99
Completed | 99
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cardiac Catheterization Patients
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.80 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 75
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 99

OUTCOME MEASURES:

1. Primary Outcome: Capsaicin Sensitivity
Description: Each patient will be asked to rate their discomfort at the application site based on a 10 point numerical rating scale for cutaneous discomfort, ranging from 0 ("no discomfort") to 10 ("the worst discomfort imaginable")
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cardiac Catheterization Patients
Number analyzed (Participants) | 98
score on a scale | 2.47 (2.15)

2. Secondary Outcome: Chest Pain Score During PCI
Description: patients are asked to rate their chest pain on a scale of 0-10 (0 "no pain", 10 "worst pain imaginable") during balloon inflation during PCI
Time Frame: approximately 1 hour
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cardiac Catheterization Patients
Number analyzed (Participants) | 98
score on a scale | 2.90 (2.92)

ADVERSE EVENTS:
Arm/Group | Cardiac Catheterization Patients
All-Cause Mortality (participants affected / at risk) | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes